CLINICAL TRIAL: NCT01907815
Title: A Phase 2 Study of MEK 1/2 Inhibitor Trametinib in Combination With AKT Inhibitor GSK2141795 in Acute Myeloid Leukemia (AML) With RAS Mutations
Brief Title: Trametinib and Akt Inhibitor GSK2141795 in Treating Patients With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01354; NCI-2013-01354 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI 9443; 2013-0001 (Other: MD Anderson Cancer Center); 9443 (Other: CTEP); N01CM39 (Other Grant/Funding Number: Federal Funding, NIH); N01CM71 (Other Grant/Funding Number: Federal Funding, NIH); P30CA016672 (NIH)
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Recurrent Adult Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — GSK2141795; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (trametinib, Akt inhibitor GSK2141795) (Experimental): Trametinib orally once daily (PO QD) and Akt inhibitor GSK2141795 PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor GSK2141795; Other: Laboratory Biomarker Analysis; Drug: Trametinib

INTERVENTIONS:
Drug: Akt Inhibitor GSK2141795 — Given PO
  Other Names: GSK2141795; Oral Akt Inhibitor GSK2141795
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist

SUMMARY:
This phase II trial studies how well trametinib and protein kinase B (Akt) inhibitor GSK2141795 work in treating patients with acute myeloid leukemia. Trametinib and Akt inhibitor GSK2141795 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the proportion of patients achieving complete remission (CR) or CR with incomplete recovery of platelets (CRp) as best response within 4 cycles of therapy of trametinib in combination with GSK2141795 (Akt inhibitor GSK2141795) in acute myeloid leukemia (AML) patients with rat sarcoma (RAS) mutations.

SECONDARY OBJECTIVES:

I. To determine the disease-free survival of patients achieving CR/CRp. II. To determine the duration of response of patients achieving CR/CRp. III. To determine the toxicity profile of trametinib in combination with GSK2141795 in this patient population.

IV. To determine the biologic effects of trametinib in combination with GSK2141795 on leukemia cells.

OUTLINE:

Patients receive trametinib orally (PO) once daily (QD) and Akt inhibitor GSK2141795 PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed AML, other than acute promyelocytic leukemia, as defined by the 2008 World Health Organization (WHO) criteria that have relapsed or refractory to standard chemotherapy; unsuitable for standard chemotherapy or unwilling to undergo standard chemotherapy; subjects >= 60 years of age with newly diagnosed AML who are not candidates for or have refused standard chemotherapy are eligible
* Patients with prior autologous and allogeneic hematopoietic stem cell transplantation are eligible if patients are off immunosuppression for > 1 month and have no evidence of active graft versus host disease (GVHD) except grade 1 skin GVHD
* Positive for RAS mutation (neuroblastoma RAS viral [v-ras] oncogene homolog [NRAS] codon 12, 13, 61 mutation or Kirsten rat sarcoma viral oncogene homolog [KRAS] codon 12, 13, 61 mutation) at a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory prior to study entry; mutational testing will be performed on bone marrow sample and/or peripheral blood; patients with previously known RAS mutations prior to study entry may be considered positive for RAS mutation for eligibility prior to a CLIA-certified laboratory confirmation of such a mutation at the discretion of the investigator; (appropriate blood and/or bone marrow samples must be taken for RAS determination and submitted to a CLIA-certified laboratory prior to study entry); however, if such a mutation is not confirmed by the M D Anderson Cancer Center (MDACC)/other center's CLIA-certified laboratory, the patient may be permitted to stay on the study if they wish and consent to do so but such patients' data will be analyzed separately
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 4 weeks
* Able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events (CTCAE) version (v)4 grade =< 1 (except alopecia) prior to the first dose of the study drug
* Serum total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (isolated total bilirubin > 1.5 institutional ULN is acceptable if bilirubin is fractionated and direct bilirubin is < 35%)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional ULN
* Serum creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) >= 60 mL/min
* Fasting serum glucose =< 150 mg/dl (fasting is defined as at least 8 hours without oral intake)
* Left ventricular ejection fraction (LVEF) >= institutional lower limit of normal (LLN) AND at least 50%; LVEF can be assessed by either echocardiogram (ECHO) or multi gated acquisition scan (MUGA)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the study participation, and for four months after the last dose of drug; women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to randomization and agree to use effective contraception throughout the treatment period and for 4 months after the last dose of study treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of another malignancy; exception: patients who have been disease-free for 3 years, or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent secondary malignancies, are eligible; consult the Cancer Therapy Evaluation Program (CTEP) Medical Monitor if unsure whether second malignancies meet the requirements specified above
* History of interstitial lung disease or pneumonitis
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to randomization; daily or weekly chemotherapy (with the exception of hydroxyurea) without the potential for delayed toxicity within 14 days prior to randomization unless there is evidence of rapidly progressive disease
* Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of trametinib/GSK2141795 and during the study
* Symptomatic or untreated leptomeningeal disease or brain metastases or spinal cord compression
* Patients with abnormal fasting glucose values (> 150 mg/dl) at screening will be excluded; in addition, patients with type 1 diabetes will also be excluded; however, patients with type 2 diabetes will be allowed if diagnosed >= 6 months prior to enrollment, and if presenting with regular hemoglobin A1C (HbA1C) =< 8% at screening
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib or excipients or to dimethyl sulfoxide (DMSO) or GSK2141795
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Other anti-cancer therapy while on study treatment; (Note: megestrol [Megace] if used as an appetite stimulant is allowed)
  * Concurrent treatment with bisphosphonates is permitted; however, treatment must be initiated prior to the first dose of study therapy; prophylactic use of bisphosphonates in patients without bone disease is not permitted, except for the treatment of osteoporosis
  * The concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's wort, kava, ephedra [ma huang], gingko biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)

    * Note: for proliferative disease, hydroxyurea will be allowed during weeks 1 and 2 of cycle 1 of study; hydroxyurea may be started or the dose changed during that 2-week period if it is clinically indicated; if a subject not previously on a stable dose of hydroxyurea needs to begin hydroxyurea or a subject on a stable dose needs to have their dose increased during the first 2 weeks, the investigator will notify the clinical team that this has been initiated
* Drugs that potently inhibit cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) should either be prohibited or used with caution; drugs which are strong inducers of cytochrome P450 family 3, subfamily A (CYP3A) should also be prohibited; drugs that are substrates of CYP3A4 or cytochrome P450 family 2, subfamily C, polypeptide 8 (CYP2C8) with a narrow therapeutic index may be prohibited; drugs that are sensitive substrates of CYP3A4 or CYP2C8 should be used with caution; it is important to regularly consult a frequently-updated list; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* History or current evidence/risk of retinal vein occlusion (RVO)
* History or evidence of cardiovascular risk including any of the following:

  * LVEF < institutional LLN or < 50%
  * A QT interval corrected for heart rate using the Bazett's formula QTcB >= 480 msec
  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to randomization are eligible)
  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to study dose are eligible)
  * Patient with symptomatic bradycardia, or a history of clinically significant bradyarrhythmias such as sick sinus syndrome, second (2nd) degree atrioventricular (AV) block (Mobitz type 2)
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to study dose
  * History or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
  * Patients with intra-cardiac defibrillators
  * Known cardiac metastases
* Known active hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (patients with chronic or cleared HBV and HCV infection, are eligible); patients with human immunodeficiency virus (HIV) are not eligible if on anti-retroviral medications
* Any serious/and or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures
* The study drug must not be administered to pregnant women or nursing mothers; women of childbearing potential should be advised to avoid pregnancy and use effective methods of contraception; men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception; if a female patient or a female partner of a patient becomes pregnant while the patient receives trametinib/GSK2141795, the potential hazard to the fetus should be explained to the patient and partner (as applicable)
* HIV-positive patients on combination antiretroviral therapy are ineligible
* Hypoxia (oxygen saturation < 90% on room air) or in the opinion of the investigator any pulmonary compromise leading to hypoxia, at the time of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 9, 2013 to January 25, 2016. All recruitment done within medical clinic settings at The University of Texas MD Anderson Cancer Center, The University of Chicago and The University of Maryland Greenebaum Cancer Center.
Pre-assignment Details: Study was terminated early, stopped due to lack of efficacy.
Groups:
- Trametinib 2.0 mg + GSK2141795 25 mg: Trametinib 2.0 mg orally once daily (PO QD) and Akt inhibitor GSK2141795 25 mg PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity
- Trametinib 1.5 mg + GSK2141795 50 mg: Trametinib 1.5 mg PO QD + GSK2141795 50 mg PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | Trametinib 2.0 mg + GSK2141795 25 mg | Trametinib 1.5 mg + GSK2141795 50 mg
Started | 17 | 7
Completed | 16 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant withdrew prior to treatment so is included in baseline demographics but not in study analysis.
Groups:
- Trametinib 2.0 mg + GSK2141795 25 mg: Trametinib 2.0 mg PO QD + GSK2141795 25 mg PO QD on days 1-28.
- Trametinib 1.5 mg + GSK2141795 50 mg: Trametinib 1.5 mg PO QD + GSK2141795 50 mg PO QD on days 1-28.
- Total: Total of all reporting groups
Arm/Group | Trametinib 2.0 mg + GSK2141795 25 mg | Trametinib 1.5 mg + GSK2141795 50 mg | Total
Number analyzed (Participants) | 17 | 7 | 24
Age, Continuous [Median (Full Range); unit: years] | 68 [22 to 80] | 69 [61 to 80] | 69 [22 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 11 | 4 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 7 | 24

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CRR, Defined as CR+CRp) Assessed by AML 2003 Response Criteria
Description: Proportion of participants achieving complete remission (CR) or CR with incomplete recovery of platelets (CRp) as best response within 4 cycles of therapy. Complete Response (CR): Disappearance all clinical &/or radiologic evidence of disease. Neutrophil count ≥ 1.0x10^9/L; Platelet count ≥ 100x109/L; Normal bone marrow differential (≤ 5% blasts); No extra-medullary leukemia. Complete Remission without Platelet Recovery (CRp): Peripheral blood & bone marrow results as for CR, but platelet counts of < 100x10^9/L. Partial Remission (PR): Blood count recovery as for CR, but decrease of at least 50% in % marrow blasts to >5% to 25% in bone marrow aspirate. Morphologic leukemia-free state: Normal marrow differential (<5% blasts); neutrophil & platelet counts not considered.95% confidence interval will be estimated for the combination regimen.
Time Frame: First four cycles (16 weeks) of therapy, with evaluation after one full cycle of therapy (28 days) and up to 16 weeks for response
Population: One participant in first cohort withdrew prior to treatment therefore excluded from study analysis.
Measure: Number; unit: percentage of participants
Groups:
- Trametinib 2.0 mg + GSK2141795 25 mg: Trametinib 2.0 mg PO QD & GSK2141795 25 mg PO QD on days 1-28.
Arm/Group | Trametinib 2.0 mg + GSK2141795 25 mg | Trametinib 1.5 mg + GSK2141795 50 mg
Number analyzed (Participants) | 16 | 7
percentage of participants | 0 | 0

2. Secondary Outcome: Most Frequently Reported Adverse Events (AE)
Description: National Cancer Institute (NCI) published standardized definitions for adverse events (AEs), known as Common Terminology Criteria for Adverse Events (CTCAE), to describe the severity of organ toxicity for those receiving cancer therapy. Toxicity data is summarized by number of incidents experienced while participants were on study using most frequently reported AEs regardless of grade or relatedness as assessed by CTCAE version 4.0. Toxicity is graded as mild (Grade 1), moderate (Grade 2), severe (Grade 3), or life-threatening (Grade 4), with specific parameters according to the organ system involved. Death (Grade 5) is used for some of the criteria to denote a fatality. For full adverse event reporting see Adverse Event Section. Data collection over first four cycles (16 weeks) of therapy, with evaluation after full cycle of therapy (28 days), continuing AE collection until 28 days following last study drug dose.
Time Frame: AE collected continuously over 28-day cycles and up to 28 days after last dose of study drug.
Population: One participant of the 17 registered in first cohort (Trametinib 2.0) withdrew without treatment and is excluded from adverse event reporting.
Measure: Number; unit: events
Groups:
- Trametinib 2.0 + GSK2141795 25 mg: Trametinib 2.0 mg PO QD + GSK2141795 25 mg PO QD on days 1-28.
Arm/Group | Trametinib 2.0 + GSK2141795 25 mg | Trametinib 1.5 mg + GSK2141795 50 mg
Number analyzed (Participants) | 16 | 7
events
  Anemia | 15 | 3
  Diarrhea | 16 | 3
  Fatigue | 11 | 6
  Fever | 13 | 3
  Nausea | 8 | 3
  Rash maculo-papular | 6 | 5
  Mucositis oral | 5 | 3
  Vomiting | 7 | 1

3. Secondary Outcome: Overall Survival of Participants Achieving CR/CRp
Description: Estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in time-to-event distributions between patient groups. Cox proportional hazards model will be used to include multiple covariates in the time-to-event analysis.
Time Frame: Up to 12 weeks
Population: No participants achieved CR/CRp therefore analysis not available.
Arm/Group | Trametinib 2.0 mg + GSK2141795 25 mg | Trametinib 1.5 mg + GSK2141795 50 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression Free Survival of Participants Achieving CR/CRp
Description: Estimated disease-free survival period using the Kaplan-Meier method. Log-rank test will be performed to test the difference in time-to-event distributions between patient groups. Cox proportional hazards model will be used to include multiple covariates in the time-to-event analysis.
Time Frame: Up to 12 weeks
Population: No participants achieved CR/CRp therefore analysis not available.
Arm/Group | Trametinib 2.0 mg + GSK2141795 25 mg | Trametinib 1.5 mg + GSK2141795 50 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Progression for Participants Achieving CR/CRp
Description: Time to Progression (TTP) is defined as the length of time from the start of treatment to disease progression as measured in days for participants with complete response.
Time Frame: Up to 12 weeks
Population: Outcome data were not collected and the Outcome will never be analyzed.
Arm/Group | Trametinib 2.0 + GSK2141795 25 mg | Trametinib 1.5 mg + GSK2141795 50 mg
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Maximum Percentage Change in Total and Phospho-proteins
Description: Change in total and phospho-proteins assessed by densitometric quantitative data by western blot analysis, or mean fluorescent intensities by flow cytometry and will be assessed for each patient for all time points and graphically plotted for each dose level.
Time Frame: Baseline to 12 weeks post therapy
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Percentage Change in Cellular Proteins
Description: The 95% confidence interval will be assessed.
Time Frame: Baseline to day 28 post treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events collected continuously over a 28-day cycle schedule and up to 28 days after last dose of study drug.
Description: One participant in first cohort withdrew prior to treatment therefore excluded from all study analysis.
Arm/Group | Trametinib 2.0 mg + GSK2141795 25 mg | Trametinib 1.5 mg + GSK2141795 50 mg
Serious Adverse Events (participants affected / at risk) | 11/16 | 6/7
Other Adverse Events (participants affected / at risk) | 16/16 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trametinib 2.0 mg + GSK2141795 25 mg (N=16) | Trametinib 1.5 mg + GSK2141795 50 mg (N=7)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Carotid Stent placed (Cardiac disorders) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Death NOS (General disorders) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspnea (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Fever (General disorders) | 2 (5) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (4) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trametinib 2.0 mg + GSK2141795 25 mg (N=16) | Trametinib 1.5 mg + GSK2141795 50 mg (N=7)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (3) | 1 (3)
Alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Alkaline phosphatase increased (Investigations) | 3 (3) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (15) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac disorders - Carotid Stent placed (Cardiac disorders) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (3) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (14) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspnea (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Edema limbs (General disorders) | 2 (2) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Esophageal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye disorders - (Other) (Eye disorders) | 2 (2) | 0 (0)
Eye infection (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (2)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 8 (11) | 5 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Fever (General disorders) | 5 (8) | 3 (3)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - (Other) (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hot flashes (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 3 (4) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infections and infestations - (Other) (Infections and infestations) | 2 (3) | 0 (0)
Injury, poisoning and procedural complications - (Other) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Lymphocyte count decreased (General disorders) | 3 (3) | 0 (0)
Malaise (General disorders) | 0 (0) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 4 (5) | 1 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - (Other) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 2 (2) | 2 (2)
Platelet count decreased (Investigations) | 4 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (4)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - (Other) (Renal and urinary disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (6) | 1 (1)
Weight loss (Investigations) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 3 (5) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less